CLINICAL TRIAL: NCT00588302
Title: Open-Label Pilot Investigation of Moexipril for the Treatment of Primary Biliary Cirrhosis (PBC)
Brief Title: Moexipril for Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1032-03
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Primary Biliary Cirrhosis
Keywords: primary biliary cirrhosis; ursodeoxycholic acid
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — moexipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A, 1 (Experimental): All patients received an open-label moexipril during the study period.
  Interventions: Drug: Moexipril

INTERVENTIONS:
Drug: Moexipril — Moexipril was given at a starting dose of 7.5 mg daily for 1 week to all enrolled patients. If tolerated (no clinically significant hypotension or medication associated adverse event), the daily dosage was increased to 15 mg daily at the beginning of the 2nd treatment week. Patients took moexipril orally in the morning and 1 hour prior to food intake. The target dose was maintained for the 1-year period of the study unless the development of toxicities warranted dose reduction or discontinuation.

SUMMARY:
The blockade of angiotensin II synthesis attenuates hepatic fibrosis in different experimental models of chronic liver injury. We aimed to determine the safety and efficacy of moexipril, an angiotensin-converting enzyme (ACE) inhibitor, on liver biochemistries, Mayo risk score, and health-related quality of life in patients with primary biliary cirrhosis (PBC) who have had a suboptimal response to ursodeoxycholic acid (UDCA).

DETAILED DESCRIPTION:
Primary biliary cirrhosis (PBC) is a chronic cholestatic liver disease of presumed autoimmune cause characterized by progressive inflammatory destruction of interlobular and septal bile ducts, resulting in fibrosis and eventual cirrhosis (1). In PBC patients, the most disabling symptoms are fatigue and pruritus which diminish health-related quality of life (HRQL. Ursodeoxycholic acid (UDCA), at a dose of 13 to 15 mg/kg per day, is a safe and effective medical therapy for most patients with PBC. Nevertheless, UDCA therapy has not ameliorated symptoms associated with PBC. Some UDCA-treated patients show progressive disease resulting in the liver transplantation or death from liver-related causes. For these patients, who show a persistent elevation of serum alkaline phosphatase at least twice the normal level after 6 months of UDCA monotherapy (incomplete responders), the evaluation of combination therapy in clinical trials has been recommended.

Moexipril is a long-acting, nonsulfhydryl ACE inhibitor with lipophilicity, and so can readily penetrate lipid membranes and thus target tissue ACE in addition to plasma ACE. This drug also demonstrated antioxidative properties in addition to efficiently controlling blood pressure in hypertensive postmenopausal subjects. Moreover, quality-of-life data suggest favorable effects of moexipril treatment in a patient population at high cardiovascular risk. The tolerability and safety profile of moexipril resembles that of other ACE inhibitors along with no reports of hepatotoxicity in controlled trials. Hence, moexipril is an attractive drug for evaluation in patients with chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* PBC patients treated with UDCA (daily dose of 13 to 15 mg/kg for at least 6 months) and an incomplete response defined by persistent elevation of serum alkaline phosphatase activity at least 2 times the upper limit of normal

Exclusion Criteria:

* age less than 18 years
* pregnancy or nursing
* anticipated need for liver transplantation within 1 year with less than a 80% one-year survival determined by the Mayo risk score
* complications of cirrhosis such as recurrent variceal hemorrhage, portosystemic encephalopathy, and refractory ascites
* history of coexistent severe cardiovascular disease including aortic stenosis
* history of coexistent severe renal disease (defined as elevation of serum creatinine more than 1.5 mg/dL) including renal artery stenosis
* history of allergy to ACE inhibitors
* current use of an ACE inhibitors or AT1 receptor antagonists in the past 3 months
* previous treatment with immunosuppressive agents or any experimental drug in the preceding 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
change in liver biochemistries and Mayo risk score for PBC | 12 months

SECONDARY OUTCOMES:
change in health-related quality of life in PBC | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Keith D Lindor, MD, Principal Investigator — Mayo Clinic and Foundation
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Talwalkar JA, Lindor KD. Primary biliary cirrhosis. Lancet. 2003 Jul 5;362(9377):53-61. doi: 10.1016/S0140-6736(03)13808-1. PMID 12853201